CLINICAL TRIAL: NCT07365631
Title: The Role of Nerve Ultrasound in Distinguishing Acquired and Genetic Sensory Neuronopathies (Ganglionopathy): A Multicenter Retrospective Study
Brief Title: Nerve Ultrasound in Acquired and Genetic Sensory Neuronopathies
Acronym: GANECHO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251638
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Sensory Neuronopathy
Keywords: Nerve ultrasound; sensory neuronopathy; ganglionopathy; CANVAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sensory neuronopathies (also called sensory ganglionopathies) are rare and heterogeneous disorders of genetic or acquired origin, caused by degeneration of the dorsal root ganglia. Their diagnosis currently relies on a combination of clinical evaluation and electrophysiological testing, as no specific biomarker is available.

Early diagnosis is particularly important in acquired forms, where early treatment can significantly influence prognosis.

Recent studies have reported a characteristic ultrasound pattern in several genetic sensory neuronopathies, showing abnormally small-caliber peripheral nerves in the upper limbs. However, these findings have only been described in genetic conditions. It is therefore unknown whether this ultrasound pattern is specific to genetic causes or may also occur in acquired sensory neuronopathies, especially those with long-standing evolution.

This retrospective multicenter study will analyze data already collected as part of routine care in approximately 50 patients with sensory neuronopathy. The objective is to compare nerve ultrasound findings between genetic and acquired forms, and to evaluate their association with clinical severity and electrophysiological parameters. Determining whether nerve atrophy observed on ultrasound is specific to genetic etiologies could help integrate ultrasound into the diagnostic workup, guiding the choice of complementary tests such as genetic analyses or early treatment initiation in acquired cases.

DETAILED DESCRIPTION:
Sensory neuronopathies (also known as sensory ganglionopathies) constitute a rare and heterogeneous group of acquired and genetic disorders related to degeneration of the dorsal root ganglia. Diagnosis relies on clinical and electrophysiological features demonstrating a pure, non-length-dependent sensory involvement. At present, no specific biomarker exists, and diagnosis is based on a combination of clinical and electrophysiological criteria. Because sensory neuronopathies are disabling conditions, early diagnosis is crucial, particularly in acquired forms for which early treatment is an important prognostic factor.

Recently, several studies have reported a unique nerve ultrasound pattern in genetic sensory neuronopathies, showing reduced caliber of mixed peripheral nerves in the upper limbs. A recent literature review suggested that sufficient evidence exists to consider ultrasound as a potential marker of genetic sensory neuronopathies. However, these studies included only patients with genetic etiologies, and no data are currently available regarding ultrasound findings in acquired sensory neuronopathies. Distinguishing between acquired and genetic causes is nevertheless essential, as the prognoses are very different and treatment must be initiated rapidly in acquired forms. Clinical evaluation alone is often insufficient to differentiate these etiologies due to substantial overlap between presentations.

The objective of this study is to compare nerve ultrasound findings in a retrospective, multicenter cohort of patients with sensory neuronopathies of either genetic or acquired origin. The study also aims to analyze correlations between nerve caliber, clinical severity, disease duration, and electrophysiological parameters. Ultimately, this research seeks to determine whether the pattern of nerve atrophy observed on ultrasound is specific to genetic causes or may also be present in acquired forms.

ELIGIBILITY:
Inclusion Criteria:

* Sensory ganglionopathy diagnosed according to the criteria of Camdessanché et al.
* Nerve ultrasound performed as part of routine clinical care.
* Age > 18 years.

Exclusion Criteria:

* Comorbid conditions that may interfere with the interpretation of sensory ganglionopathy.
* Lack of consent (patient opposition to the use of clinical data for research).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with sensory neuronopathy according to Camdessanché criteria, who underwent nerve ultrasound as part of routine clinical care. Patients are retrospectively identified from medical records across four French tertiary neurology centers between 2024 and 2025, including both acquired and genetic etiologies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area of peripheral nerves according to ganglionopathy etiology (genetic vs acquired) | Baseline
  Measurement of the cross-sectional area (mm²) of peripheral nerves on ultrasound (median nerve at forearm and arm, ulnar nerve at forearm and arm, sural nerve at ankle, radial sensory nerve at distal forearm, C5 and C6 roots at foraminal emergence, and vagus nerve at mid-cervical level) to compare nerve caliber between patients with genetic versus acquired sensory ganglionopathies

SECONDARY OUTCOMES:
Correlation between nerve cross-sectional area and clinical severity | Baseline
  Assessment of the association between peripheral nerve cross-sectional area (mm²) and clinical variables, including duration of symptoms (months) and severity of proprioceptive ataxia (Mariette score, 0-3)
Correlation between nerve cross-sectional area and electrophysiological severity | Baseline
  Assessment of the association between peripheral nerve cross-sectional area (mm²) and electrophysiological parameters, including sensory nerve action potential amplitudes (sural and radial nerves, µV) and other available electrophysiological measures relevant to axonal loss

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FARGEOT, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris